CLINICAL TRIAL: NCT04044391
Title: Noninvasive Magnetocardiography Using the CardioFlux (TM) System in the Evaluation of Acute Coronary Syndrome Patients Going for Cardiac Catheterization
Brief Title: Use of Magnetocardiography in Evaluation of Patients Going for Cardiac Catheterization
Status: Terminated | Type: Observational
Why Stopped: Study was defunded.
Sponsor: Genetesis Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1345773
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Acute Coronary Syndrome; Coronary Artery Stenosis; Myocardial Ischemia
Keywords: Coronary Artery Disease; Myocardial ischemia
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Stenosis; Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Intention to Treat: Cardiac Catheterization: All patients meeting inclusion criteria and scheduled to undergo cardiac catheterization will undergo a CardioFlux magnetocardiogram (MCG) to determine presence of patterns which indicate myocardial ischemia.
  Interventions: Diagnostic Test: CardioFlux Magnetocardiograph
- Post Percutaneous Coronary Intervention: All patients found to have significant coronary artery obstruction seen via angiography +/- fractional flow reserve (FFR) or instant wave-free ratio (iFR) and who receive a catheter based intervention will have a post-procedure CardioFlux MCG scan. Follow up over the next 30 and 180 days will be performed to determine if a persistent pattern suggesting residual ischemia will correlate with an increased incidence of major cardiac adverse events (MACE).
  Interventions: Diagnostic Test: CardioFlux Magnetocardiograph

INTERVENTIONS:
Diagnostic Test: CardioFlux Magnetocardiograph — CardioFlux is a noninvasive diagnostic modality which can measure and image the heart's intrinsic magnetic field created by ion transit across cardiac cell membranes.

SUMMARY:
This is a multicenter, prospective trial to measure the test performance characteristics of the Magnetocardiography (MCG) CardioFlux cardiac diagnostic system in detecting clinically significant coronary artery obstruction in patients with symptoms of suspected acute coronary syndrome or who present with a failed stress test with the intention of treat with cardiac catheterization.

DETAILED DESCRIPTION:
This is a multicenter, prospective clinical trial studying the utility and accuracy of magnetocardiography (MCG) in identifying critical coronary artery obstruction responsible for myocardial ischemia. The study will enroll up to 1500 patients at high risk for coronary artery disease (CAD) who have been referred for cardiac catheterization. These patients will be recruited from an inpatient service post admission for chest pain or anginal equivalent or from a cohort of symptomatic patients who have failed outpatient stress testing. If they meet other stated inclusion criteria, they will have a 2 minute MCG scan prior to their cardiac catheterization. For comparative purposes, the first 300 patients will have an electrocardiogram (ECG) performed within 60 minutes of this initial scan.

After an enrolled study subject has had their catheterization procedure, the results of the catheterization will be reviewed by one of the study's primary investigators. If the subject has had a percutaneous coronary intervention (PCI), a second MCG scan will be performed prior to their discharge. The MCG scans will be interpreted by 3 physicians trained to read these images and blinded to all clinical information regarding study subjects.

The initial MCG scan will be evaluated for its sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and overall accuracy in detecting myocardial ischemia and critical coronary stenosis based on angiographic imaging, fractional flow reserve (FFR), or instant wave-free ratio (iFR) measurements, as applicable. The same statistical analysis will be performed for the ECGs performed on each of the applicable study subjects. When performed, the second MCG will be evaluated for any abnormalities after revascularization. These results will be used to determine the value of post-PCI MCG to predict 30 day and 180 day major adverse cardiac events (MACE)-specifically myocardial infarction or stroke, need for revascularization, or cardiac related death.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age at the time of enrollment.
* Patient presenting acutely with signs and symptoms suggestive of Acute Coronary Syndrome (ACS) and in the opinion of the treating physician and based on best clinical assessment that a cardiac catheterization will be performed; or, had a positive stress test and is scheduled for cardiac catheterization.
* Patient's ability to lay supine for five minutes.

Exclusion Criteria:

* Age < 18 years of age
* Patients unable to fit into device
* Unable to transfer to device gantry
* Positive response on magnetocardiography (MCG) prescreening form
* Patients with claustrophobia or unable to lie supine for five minutes
* Pregnant women
* Poor candidate for follow-up (e.g. no access to phone)
* Repeat participants
* Prisoners
* Acute STEMI or hemodynamically unstable patients (Mean Arterial Pressure ≤ 65, Respiratory Rate ≥24, Heart Rate ≥105 bpm, Temperature>38.1 or <34 degrees Celsius, O2 Saturation<90% despite oxygen therapy).
* Do not resuscitate order (DNR)
* Unable to have a cardiac catheterization secondary to dye, allergy, creatinine clearance, can't obtain access, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This research study will enroll patients who will undergo cardiac catheterization because of symptoms and risk factors suggestive of acute coronary syndrome, and high risk patients presenting for cardiac catheterization due to an abnormal stress test. Patients meeting these criteria, and over the age of 18 years and all genders will be candidates.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Accuracy of MCG to detect myocardial ischemia as determined by cardiac catheterization | 72 hours
  Assess accuracy of CardioFlux MCG (MCG-CF) and magnetic field map characteristics with findings of significant coronary artery stenosis ≥70% via angiography and/or via FFR of <0.8 or via instant wave-free ratio (iFR) .
Accuracy of MCG vs. ECG | 72 hours
  Compare CardioFlux MCG accuracy to ECG accuracy in identifying cardiac ischemia using coronary angiography with or without FFR/iFR as gold standard.

SECONDARY OUTCOMES:
Incident of post-PCI MACE | 6 months
  Determine if residual abnormalities on post PCI MCG-CF maps can predict 30 day and 180 day MACE.
Inter-reader reliability percentage | 6 months
  Measurement of consistency of interpretation among 3 physician readers of CardioFlux MCG scans.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Pearson, M.D., Principal Investigator — Ascension St, John Medical Center
Locations (2):
- United States (2):
  - Ascension St. John Medical Center, Detroit, Michigan
  - Beaumont Hospital, Royal Oak, Michigan

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual patient data (IPD) available to researchers not affiliated with the centers enrolling patients within this trial.

REFERENCES:
- [Background] Chaikovsky I, Hailer B, Sosnytskyy V, Lutay M, Mjasnikov G, Kazmirchuk A, Bydnyk M, Lomakovskyy A, Sosnytskaja T. Predictive value of the complex magnetocardiographic index in patients with intermediate pretest probability of chronic coronary artery disease: results of a two-center study. Coron Artery Dis. 2014 Sep;25(6):474-84. doi: 10.1097/MCA.0000000000000107. PMID 24667125
- [Background] Chen T, Z., C., Jiang, S, Van Leeuwen, P., Gronemeyer, D, Noninvasively diagnosing coronary artery disease with 61 channel MCG data. Chinese Science Bulletin. , 2014. 59: p. 1123.
- [Background] Hailer B, Chaikovsky I, Auth-Eisernitz S, Schafer H, Van Leeuwen P. The value of magnetocardiography in patients with and without relevant stenoses of the coronary arteries using an unshielded system. Pacing Clin Electrophysiol. 2005 Jan;28(1):8-16. doi: 10.1111/j.1540-8159.2005.09318.x. PMID 15660796
- [Background] Park JW, Hill PM, Chung N, Hugenholtz PG, Jung F. Magnetocardiography predicts coronary artery disease in patients with acute chest pain. Ann Noninvasive Electrocardiol. 2005 Jul;10(3):312-23. doi: 10.1111/j.1542-474X.2005.00634.x. PMID 16029382
- [Background] Lim HK, Kwon H, Chung N, Ko YG, Kim JM, Kim IS, Park YK. Usefulness of magnetocardiogram to detect unstable angina pectoris and non-ST elevation myocardial infarction. Am J Cardiol. 2009 Feb 15;103(4):448-54. doi: 10.1016/j.amjcard.2008.10.013. Epub 2008 Dec 25. PMID 19195500
- [Background] Li Y, Che Z, Quan W, Yuan R, Shen Y, Liu Z, Wang W, Jin H, Lu G. Diagnostic outcomes of magnetocardiography in patients with coronary artery disease. Int J Clin Exp Med. 2015 Feb 15;8(2):2441-6. eCollection 2015. PMID 25932186
- [Background] Kwong JS, Leithauser B, Park JW, Yu CM. Diagnostic value of magnetocardiography in coronary artery disease and cardiac arrhythmias: a review of clinical data. Int J Cardiol. 2013 Sep 1;167(5):1835-42. doi: 10.1016/j.ijcard.2012.12.056. Epub 2013 Jan 19. PMID 23336954
- [Background] Agarwal R, Saini A, Alyousef T, Umscheid CA. Magnetocardiography for the diagnosis of coronary artery disease: a systematic review and meta-analysis. Ann Noninvasive Electrocardiol. 2012 Oct;17(4):291-8. doi: 10.1111/j.1542-474X.2012.00538.x. Epub 2012 Aug 13. PMID 23094875
- [Background] Kwon H, Kim K, Lee YH, Kim JM, Yu KK, Chung N, Ko YG. Non-invasive magnetocardiography for the early diagnosis of coronary artery disease in patients presenting with acute chest pain. Circ J. 2010 Jul;74(7):1424-30. doi: 10.1253/circj.cj-09-0975. Epub 2010 May 27. PMID 20508380
- [Background] Tolstrup K, Madsen BE, Ruiz JA, Greenwood SD, Camacho J, Siegel RJ, Gertzen HC, Park JW, Smars PA. Non-invasive resting magnetocardiographic imaging for the rapid detection of ischemia in subjects presenting with chest pain. Cardiology. 2006;106(4):270-6. doi: 10.1159/000093490. Epub 2006 May 29. PMID 16733351